CLINICAL TRIAL: NCT00590811
Title: Prevalence of Menstrual Cycle Related Pain Complains in Adolescents and Young Adults
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Christel Meuleman, MD, University Hospital Leuven, Leuven, Belgium
Other Study IDs: EC - 14/11/2007
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-01

CONDITIONS: Dysmenorrhea; Pelvic Pain
Keywords: adolescents; young adults; dysmenorrhea; pelvic pain
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- adolescents: 3rd year high school girls (14-16 years old)
- young adults: 1st year university young females (18 - 20 years old)

SUMMARY:
The aim of this study is to determine the prevalence of menstrual cycle related pain complains in adolescents and young adults.

DETAILED DESCRIPTION:
An internet questionnaire with 12 items was used:

Adolescents

* start of menstruation
* characteristics of menstrual cycle
* pain related to menstrual cycle (questions based on well-known pain-complaints related to the presence of endometriosis)
* analgetics
* influence on school carrier
* influence on social life

Young adults

* idem as for adolescents
* influence of pain on an eventual sexual relationship

ELIGIBILITY:
Inclusion Criteria:

* 3rd year high school girls
* 1st year university young females

Exclusion Criteria:

* pre-menarcheal girls

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 3rd year high school girls and 1st year university young females having a routine visit to the school doctor or student doctor.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of menstrual cycle related pain complains | 3rd year high school & first year university

SECONDARY OUTCOMES:
Relationship between level of pain complains and characteristics of menstrual cycle | 3rd year high school & first year university

CONTACTS AND LOCATIONS:
Overall Officials: Christel LC Meuleman, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (2):
- Belgium (2):
  - MPTC, Leuven
  - VCLB, Leuven